CLINICAL TRIAL: NCT02476240
Title: Can Dual Task Walking Improve in Parkinson's Disease After External Focus of Attention Exercise? A Single Blind Randomized Controlled Trial
Brief Title: Evaluating the Influence of Externally vs. Internally Focused Exercise on Rehabilitation in Parkinson's Disease
Acronym: DT-PDSAFEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Eric Beck, Graduate Student, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3983
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease
Keywords: Exercise; Attention
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Internally Focused PD-SAFEx (Active Comparator): While performing the exercises in PD-SAFEx™, participants will be instructed to focus their attention on sensory feedback. This will include focusing participants' attention on the stretch in their limbs while walking, on the straightness of their backs while sitting, on limb and body orientation in space while coordinating their movements, and on chest movements during breathing exercises. Throughout each exercise session, the instructor and volunteers will constantly provide attention-directing instructions.
  Interventions: Behavioral: Parkinson's disease Sensory Attention Focused Exercise
- Externally Focused PD-SAFEx (Experimental): While performing the exercises from the PD-SAFEx™ program, participants will be instructed to focus their attention externally on the movement of coloured labels attached to their feet, knees, elbows and hands. Participants will be reminded and encouraged by the exercise instructor and volunteers to perform all exercises while focusing attention on the labels.
  Interventions: Behavioral: Parkinson's disease Sensory Attention Focused Exercise
- Control Group (No Intervention): This group will be asked to refrain from changing activities of their daily lives throughout the 20-week duration of the experiment (from pre-assessment to washout).

INTERVENTIONS:
Behavioral: Parkinson's disease Sensory Attention Focused Exercise — The first half of the exercise class will include walking exercises that include large magnitude and coordinated movements. All walking will be performed slowly. Walking exercises will be followed by balance, stretching, and coordination exercises while sitting in, or standing near, standard office chairs, utilizing latex Thera-bands®. To ensure that balance and coordination are constantly challenged throughout the intervention, the exercise program progresses each week, increasing in difficulty. Depending on the task, the first set of each exercise will be performed with 'eyes-open' to familiarize participants with the task, and subsequent sets will be performed with 'eyes-closed'. If there is only one set for a specific exercise, the first half of the repetitions will be performed with 'eyes-open' and the second half with 'eyes-closed'.
  Other Names: PD-SAFEx
  Arms: Externally Focused PD-SAFEx; Internally Focused PD-SAFEx

SUMMARY:
The purpose of this study is to evaluate the underlying mechanism and influence of externally vs. internally focused exercise on rehabilitation in Parkinson's disease. The upcoming exercise intervention methodology will aim to meet the requirements of a 1A silver ranking level, single blind, randomized control trial according to the criterion of the Cochrane Musculoskeletal Review Group

DETAILED DESCRIPTION:
Parkinson's disease is a slow progressing neurodegenerative movement disorder with both motor and non-motor symptoms. The gold standard medical pharmacotherapy (levodopa) lends relief from symptoms. However, some of the non-motor symptoms are not responsive to this therapy or eventually become non-responsive, such as impaired proprioception (sensory feedback from the limbs providing awareness of one's body in physical space). Although it is unclear as to why levodopa is unable to relieve proprioception impairments, a key underlying mechanism that may be responsible is an impaired sensorimotor integration (the combination of sensory and motor information in the brain utilized to guide movements). This is not the result of corrupted input information from proprioceptors into the brain (such as muscle spindles and golgi tendon organs), but rather the downstream integration of this information in the brain. With faulty signalling through the area of the brain damaged in Parkinson's disease (the basal ganglia), deficient sensorimotor integration impairs patients' ability to rely on sensory feedback during movement. This subsequently impairs ability to automatize learned movements in Parkinson's disease and causes previously automatic movements (such as walking) to require conscious control (lose automaticity). This is problematic in instances where attention is diverted from a movement that is no longer automatically controlled, such as engaging in a conversation while walking. Without attention on the movement, motor control breaks down, leading to heightened chance of falls and injury. However, Wulf and Colleagues (2009) demonstrated that when individuals with Parkinson's disease focused externally, and greater reliance on sensorimotor integration was fostered, balance control was improved compared to when these individuals focused attention internally. This suggests that individuals with Parkinson's disease may retain ability to rely on sensorimotor integration. Therefore, by fostering neuroplasticity through the basal ganglia with the utilization of exercise, and improving ability to rely on sensorimotor integration in individuals with Parkinson's disease (by using dual task training), automaticity of movements may be improved, subsequently decreasing the risk of falling and injury. Furthermore, by improving sensorimotor integration, symptom severity might improve and disease progression may slow.

In addition to providing improvements to symptoms of Parkinson's disease, this will provide a greater understanding into the pathophysiological mechanisms underlying improvements associated with exercise rehabilitations employed for Parkinson's disease. To date, goal-directed exercises have yet to investigate the rudimentary aspects of the exercise, since no studies have directly compared identical exercise regimens while participants focus "internally" on the movements of their limbs compared to focusing "externally" on the movement of an object that is being manipulated. For this reason, this study will investigate large magnitude gait and balance training in two groups, one focusing internally on limb movements throughout the exercise program, and the other focusing externally on the movement of coloured labels attached to their limbs. The gait, balance, stretching and coordination exercises that will be provided in the proposed intervention to the two exercise groups will follow the exact Parkinson's disease Sensory Attention Focused Exercise (PD-SAFEx™) protocol designed by Sage and Almeida (2009). PD-SAFEx™ is a group setting intervention, which will be led by the primary investigator who is trained in conducting the exercise protocol. The first half of the exercise class will include walking exercises that include large magnitude and coordinated movements. All walking will be performed slowly. Walking exercises will be followed by balance, stretching, and coordination exercises while sitting in, or standing near, standard office chairs, utilizing latex Thera-bands®. To ensure that balance and coordination are constantly challenged throughout the intervention, the exercise program progresses each week, increasing in difficulty.

Sixty-five participants diagnosed with idiopathic Parkinson's disease will be recruited. This present intervention study will span over a 20- week period. Pre-assessments to measure baseline symptoms and functionality will be conducted over the initial 2-week period prior to the start of the intervention. After pre-assessments have been conducted, participants will be randomized to one of three groups:

Group 1: Internal Focus of attention Exercise (Original PD-SAFEx™) While performing the exercises in PD-SAFEx™, participants will be instructed to focus their attention on sensory feedback. This will include focusing participants' attention on the stretch in their limbs while walking, on the straightness of their backs while sitting, on limb and body orientation in space while coordinating their movements, and on chest movements during breathing exercises. Throughout each exercise session, the instructor and volunteers will constantly provide attention-directing instructions.

Group 2: External Focus of attention Exercise (Modified PD-SAFEx™) While performing the exercises from the PD-SAFEx™ program, participants will be instructed to focus their attention towards the movement of coloured labels attached to their hands, elbows, knees and feet.

Group 3: Control Group This group will be asked to refrain from changing activities of their daily lives throughout the 20-week duration of the experiment (from pre-assessment to washout).

The exercise program will follow the pre-assessment baseline measures, and will last 12 weeks. Each exercise session will last 60 minutes, and will be provided three times per week. Post-assessment of all outcome measures tested prior to the intervention will be assessed in a 2-week period immediately after the cessation of the exercise program. The washout period will last 6 weeks; thereafter assessments will be completed again. Since the present research study aims to understand the mechanism underlying these rehabilitations, as well as ensure ecological validity, symptom severity (UPDRS-III) will be assessed in all individuals in both the "ON" and "OFF" state of dopaminergic medication. Since the individuals are in the "ON" state during all daily activities, exercise classes will be performed in the "ON" dopaminergic medication state. If there are individuals who are naïve to dopaminergic medication (De novo), they will only be assessed once (in the "OFF" dopaminergic state). All individuals included in the rehabilitation program will be required to complete a Physical Activity Readiness Medical Examination (ParMed X), signed by a physician prior to joining the rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Either gender, no age or location restriction
* Diagnosed with idiopathic Parkinson's disease by a Neurologist
* Able to stand 2 minutes, unassisted
* Able to walk 10 meters, unassisted
* Able to understand English instructions

Exclusion Criteria:

* A neurological disease other than Parkinson's disease
* Peripheral neuropathy
* Clinically diagnosed with dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease Rating Scale Part III (UPDRS-III) | Pre-assessment to post-assessment (12 weeks)
  A physical movement assessment to quantify Parkinson's disease symptom severity. This is a non-invasive, risk free, painless examination.
UPDRS-III | Post-assessment to Washout (8 weeks)
  A physical movement assessment to quantify Parkinson's disease symptom severity. This is a non-invasive, risk free, painless examination.
Single and Dual Task Walking | Pre-assessment to Post-assessment (12 weeks)
  Participants will be asked to walk along a 9.75m long and 0.61m wide ProtoKinetics Movement Analysis Software™ electronic walkway carpet (Zeno Walkway - ProtoKinetics, Havertown, PA, USA). This electronic walkway will measure spatiotemporal characteristics of the individuals' gait while they walk with and without the performance of a dual task. The dual task that will be performed by the participants with Parkinson's disease will be a phoneme monitoring dual task not trained in the intervention. Participants will be asked to complete 3 trials of each condition.
Single Task and Dual Task Walking | Post-assessment to washout (8 weeks)
  Participants will be asked to walk along a 9.75m long and 0.61m wide ProtoKinetics Movement Analysis Software™ electronic walkway carpet (Zeno Walkway - ProtoKinetics, Havertown, PA, USA). This electronic walkway will measure spatiotemporal characteristics of the individuals' gait while they walk with and without the performance of a dual task. The dual task that will be performed by the participants with Parkinson's disease will be a phoneme monitoring dual task not trained in the intervention. Participants will be asked to complete 3 trials of each condition.
Parkinson Anxiety Scale Questionnaire | Pre-assessment to Post-assessment (12 weeks)
  Valid measure of persistent, episodic, and avoidance behaviour anxiety
Parkinson Anxiety Scale Questionnaire | Post-assessment to washout (8 weeks)
  Valid measure of persistent, episodic, and avoidance behaviour anxiety

SECONDARY OUTCOMES:
Measures of Executive Function | Pre-assessment to post-assessment (12 weeks)
  To measure general cognitive status, the Montreal Cognitive Assessment will be completed.
Measures of Executive Function | Post-assessment to Washout (8 weeks)
  To measure general cognitive status, the Montreal Cognitive Assessment will be completed.
Parkinson's disease Questionnaire 39 | Pre-assessment to Post-assessment (12 weeks)
  A validated questionnaire for individuals with Parkinson's disease to address well-being and perceived quality of life.
Parkinson's disease Questionnaire 39 | Post-assessment to washout (8 weeks)
  A validated questionnaire for individuals with Parkinson's disease to address well-being and perceived quality of life.
Community Health Activities Model Program for Seniors questionnaire (CHAMPS) | Pre-assessment to post-assessment (12 weeks)
  To determine whether the control group changes in physical activity level throughout the duration of the present study
CHAMPS | Post-assessment to washout (8 weeks)
  To determine whether the control group changes in physical activity level throughout the duration of the present study

CONTACTS AND LOCATIONS:
Overall Officials: Quincy J Almeida, PhD, Study Director — Sun Life Financial Movement Disorders Research and Rehabilitation Centre, Wilfrid Laurier University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wulf G, Landers M, Lewthwaite R, Tollner T. External focus instructions reduce postural instability in individuals with Parkinson disease. Phys Ther. 2009 Feb;89(2):162-8. doi: 10.2522/ptj.20080045. Epub 2008 Dec 12. PMID 19074619
- [Background] Sage MD, Almeida QJ. Symptom and gait changes after sensory attention focused exercise vs aerobic training in Parkinson's disease. Mov Disord. 2009 Jun 15;24(8):1132-8. doi: 10.1002/mds.22469. PMID 19373930
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886